CLINICAL TRIAL: NCT00983762
Title: Comparison of Functional Outcomes of Three Surgical Approaches in Knee Arthroplasty: The Minimally Invasive Surgery Mini-Incision (MIS) TKA, Standard Para-Patellar Surgery TKA and the Unicompartmental Knee Arthroplasty
Brief Title: Comparison of Functional Outcomes of Three Surgical Approaches in Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: No continued funding.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Henrik Malchau, PhD, MD, Massachusetts General Hospital
Other Study IDs: 2007P001220
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Leg strength; Functional outcomes; Minimally Invasive Surgery Mini-Incision (MIS) TKA; Unicompartmental knee arthroplasty; Standard Para-patellar surgery TKA; gait; knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- MIS knee arthroplasty: Persons scheduled for Minimally Invasive Surgery Mini-Incision (MIS) Total Knee Arthroplasty (TKA)
- Unicompartmental knee arthroplasty: Persons scheduled for Unicompartmental knee arthroplasty
- Standard knee arthroplasty: Persons scheduled for Standard Para-patellar surgery TKA
- Heathly knee subjects: Persons with healthy knees

SUMMARY:
A functional outcomes comparison study of three surgical techniques using minimally invasive surgery mini-incision (MIS) for total knee arthroplasty (TKA), standard para-patellar TKA and the unicompartmental knee arthroplasty performed over a 2+ year post-op period.

DETAILED DESCRIPTION:
The purpose of this research study is to compare post-operative knee function of persons who have undergone one of three types of knee arthroplasty for the treatment of knee osteoarthritis. A variety of functional performance tests will be assessed and compared using a group of evaluations including: functional activity performance tests and questionnaires; leg strength; knee range of motion; and forces at the knee during a series of activities (walking, bending, stepping etc.) via a motion analysis system. The study will compare the three surgical subject groups and one group of healthy, non-surgical subjects for a total of 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

* TKA subjects:

  1. Patients requiring primary knee arthroplasty;
  2. Knee osteoarthritis;
  3. Subject has sufficient quantity or quality of bone support;
  4. Subject has no previous or active infection in the affected joint or systemic infection;
  5. Subject judged to be available for follow-up through at least 1 year postoperative;
  6. All subjects in arthroplasty groups will be between 50-70 years of age
* Healthy subjects:

  1. Healthy subjects will have no complaints of knee pain or history of knee surgery or known arthritic knee changes.
  2. All subjects will have no history of prior lower extremity arthroplasty surgeries or systemic disease which could confound outcome measures.
  3. All healthy persons will be 40-70 years.

Exclusion Criteria:

1. Insufficient quantity or quality of bone support resulting from conditions such as cancer, femoral osteotomy, significant osteoporosis or metabolic disorders of calcified tissues;
2. Unable to return for follow up x-rays and clinical evaluation;
3. Unable to comprehending study protocol for any reason;
4. Systemic inflammatory joint disease (rheumatoid arthritis), previous infection or those requiring revision knee surgery;
5. Subject has an immunological disorder: immunosuppressive treatment characterized by markedly inhibited ability to respond to antigenic stimuli. Examples of such conditions include Subjects who are on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses), Subjects receiving therapy to prevent homograft rejection, Subjects who have a documented history of acquired immunodeficiency syndrome (AIDS), or auto-immune diseases;
6. Subject has a neurologic condition that would influence the results of biomechanical analysis of whole body movement.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TKA subjects:
  Subjects will be selected and recruited from the MGH Arthroplasty Clinic. The surgical decision for TKA approach will be made prior to recruitment for the study.
  Healthy persons:
  Healthy subjects will be recruited through orthopedic departmental advertisement flyers and by word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic and isometric quadriceps and hamstring strength | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years

SECONDARY OUTCOMES:
American Academy Orthopaedic Surgeons Knee Score | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
University California Los Angeles Activity Score | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Timed "Up & Go" Test | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Sit to Stand to Sit (STSTS) Test | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Stair Test | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Visual Analog Pain Scale | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Knee adductor moment during gait and chair rise | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years
Knee loading pattern during gait & chair rise | Pre-op, post op: 4 weeks, 3 months, 6 months and at 1, 2, 5, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Malchau, PhD, MD, Principal Investigator — Massachusetts General Hospital